CLINICAL TRIAL: NCT05843474
Title: Effectiveness of Take it Personal! A Substance Use Intervention for Young People With Mild Intellectual Disabilities and Borderline Intellectual Functioning
Brief Title: Effectiveness of Take it Personal!
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Behavioural Science Institute (Other)
Collaborators: Pluryn (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 555002014
Record Dates: First submitted 2023-01-16; First posted 2023-05-06 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-03

CONDITIONS: Alcohol Use; Drug Use; Mild Intellectual Disability, IQ 50-70; Borderline Intellectual Disabilities (Intelligence Quotient 70-85); Personality; Adolescent Behavior
MeSH Terms: conditions — Alcohol Drinking; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: a non-concurrent ABA multiple baseline design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Take it Personal! — Take it Personal! is a six-week indicated prevention program for youth with a mild intellectual disability or borderline intellectual functioning. The program aims to teach youngsters skills to reduce their substance use (alcohol, cannabis, and other drugs). The prevention program differentiates four personality profiles associated with a higher risk for problematic substance use: sensation seeking, impulsivity, anxiety sensitivity and negative thinking. For each of the four personality profiles, different program outlines were developed that are similar in structure but have their own personality-specific materials, games and (psychomotor) exercises. There are weekly individual- and group sessions with three to four participants, led by a clinical psychologist and a psychomotor therapist. Motivational interviewing and cognitive behavioral therapeutic principles are applied, both of which have proven effectiveness in decreasing substance use the target group.

SUMMARY:
A controlled pre-post design study on Take it Personal! has demonstrated effectiveness in reducing the frequency and severity of youth use of alcohol, cannabis or other illicit drugs. Take it Personal! is an existing indicated prevention programme for substance use in youth with a mild intellectual disability or borderline intellectual functioning that addresses each participant's high-risk personality traits for substance abuse. The current Take it Personal! programme is further developed and optimized in collaboration with relevant stakeholders. In particular, the investigators aim to integrate personalized daily diary monitoring in the programme so that trainers can monitor client progresses closely and gain insights into change mechanisms, providing starting points for therapeutic efforts in programme sessions. The investigators conduct a series of case studies with a non-concurrent multiple baseline design to evaluate the effectiveness of Take it Personal!. The baseline lengths are randomly determined, and therefore the start of the intervention is staggered across participants.

DETAILED DESCRIPTION:
Procedure Participants have either 14, 17, 20 or 23 days of baseline measurements. After baseline, participants will follow Take it Personal! for six weeks. Lastly, there is a follow-up phase in which each participant completes 30 days of daily diaries.

The Ethica mobile phone application is used for data collection, which facilitates user-friendly editing and adding of items to optimally personalize monitoring and care. Trainer and client can translate intervention goals into the participant's daily diary items. Completing daily diaries primarily has a clinical incentive for participants, as responses are discussed in Take it Personal!. That is, during the programme, data are fed back to the therapists to facilitate deeper knowledge on participant's behavioural and affective patters. In individual sessions, participant and trainer will inspect and interpret the daily monitoring data to gain more structured insights into changes over time.

To gain additional insight into the long-term effects on substance use frequency, problems caused by substance use and symptoms of dependence, the investigators administer the Alcohol Use Disorders Identification Test (AUDIT) and the Drug Use Disorders Identification Test (DUDIT), which are incorporated as subscales in the Substance Use and Misuse among Intellectually Disabled Persons Questionnaire (SumID-Q) and this survey's collateral report version (SumID-CR) to respectively participants and daily carers at baseline, 1-, 6- and 12-month follow-up.

The investigators add complementary qualitative components that will enable better interpretation of why changes occur or not occur for individuals. One month after the last Take it Personal! session, the Client Change Interview (CCI) is administered to the participant and his/her daily carer separately. The CCI is a semi structured interview, previously used in a mild intellectual disability, in which participants reflect on changes they did and did not notice since starting the programme and contemplate on what caused this. During the CCI, participant and the participant's primary carer are asked to reflect on during which periods changes occurred.

Sample size 15 participants

Sample size justification The joint Dutch quality assessment procedure ('erkenningstraject effectieve interventies') states that a series of at least 10 well-executed case studies, under different conditions and different therapists, is recognized to demonstrate strong evidence for intervention and prevention effectiveness. The investigators obtain an additional 30% to account for withdrawal, drop-out, missing data, and decreasing adherence rates, resulting in a required sample size of 15 participants who will enroll in a non-concurrent multiple baseline study with different therapists per group.

ELIGIBILITY:
Inclusion criteria:

* Between 14 and 30 years of age
* A DSM-5 based diagnosis of mild intellectual disability OR borderline intellectual functioning A mild intellectual disability is characterized by an intelligence quotient (IQ) score between 50-70 and limitations in adaptive behavior that impede a range of everyday social and practical skills. The DSM-5 describes borderline intellectual functioning as a condition in which a person's limited intellectual functioning is the focus of, or has an impact on, their treatment. This diagnosis is typically given when IQ is roughly between 70 and 85. Persons with either diagnosis often lead problematic lives, facing, for example, social and coping difficulties, and are vulnerable to the development of psychopathologies such as substance use disorder.
* Receives specialized in- or outpatient care
* Uses alcohol or drugs at least once per two weeks, as confirmed by participant's clinician
* Owns a mobile phone

Exclusion criterium

- Moderate or severe substance use disorder

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in daily substance use frequency | Through study completion, on average 90 days
  Daily diaries include at least one item about substance use. Depending on which substance the individual uses, it will inquire after units of the substance used per day. For example, "how many glasses of alcohol did you drink today?" or "how many joints did you smoke today?"

SECONDARY OUTCOMES:
Change in daily personal behavioral problem | Through study completion, on average 90 days
  Daily diaries will include at least one item about personally relevant issues that the participant wants to work on in Take it Personal! which will be rated on a 5-point Likert scale ranging from "not at all" to "very much".
Change in substance use frequency | Baseline, 1-month, 6-month, and 12-months
  Measured with SumID-Q survey at baseline, 1-month post-intervention, 6-month post-intervention, and 12-months post-intervention
Experienced changes | 1 month
  The Client Change Interview that is administered one month post-intervention. The interview maps out which behavioral changes the client noticed since starting Take it Personal!, the importance they had, and to which causes the client attributes these changes. These qualitative results are presented descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Poelen, PhD, Principal Investigator — Radboud University and Pluryn
Locations (1):
- Behavioural Science Institute, Radboud University, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Preregistration, metadata and analyses scripts/syntax will be stored in the Open Science Framework (OSF; www.osf.io) and will be made findable and accessible publicly. The raw data (i.e., pseudonymized quantitative data in .csv of daily diaries, standardized surveys and anonymized transcripts of the client change interviews), as well the metadata, will be made findable and openly accessible on the repository of Radboud University: Radboud Repository. A persistent identifier will be made through OSF, which is then also included in the Radboud Repository. Hence, we use only one DOI. Sensitive data cannot be made publicly accessible. Therefore, audio recordings of the interviews nor any contact information (names, e-mail addresses, addresses) are not accessible.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Babor, T. F., Higgins-Biddle, J. C., Saunders, J. B., & Monteiro, M. G. (2001). AUDIT. The alcohol use disorders identification test. Guidelines for use in primary care. Geneva: World Health Organisation.
- [Background] Berman, A. H., Bergman, H., Palmstierna, T., & Schlyter, F. (2003). DUDIT. The drug use identification test manual. Stockholm: Karolinska Institutet, department of clinical neuroscience.
- [Background] Kazdin AE. Understanding how and why psychotherapy leads to change. Psychother Res. 2009 Jul;19(4-5):418-28. doi: 10.1080/10503300802448899. PMID 19034715
- [Background] Wieland J, Zitman FG. It is time to bring borderline intellectual functioning back into the main fold of classification systems. BJPsych Bull. 2016 Aug;40(4):204-6. doi: 10.1192/pb.bp.115.051490. PMID 27512590
- [Background] Thompson B, Tickle A, Dillon G. Discovery awareness for staff supporting individuals with intellectual disabilities and challenging behaviour: is it helpful and does it increase self-efficacy? Int J Dev Disabil. 2019 Apr 20;67(1):44-57. doi: 10.1080/20473869.2019.1599605. PMID 34141398
- [Background] Zwikker, M., van Dale, D., Dunnink, T., Willemse, G, van Rooijen, S., Heeringa, N., & Rensen, P. (2015). Erkenning van interventies. Criteria voor gezamenlijke kwaliteitsbeoordeling 2015-2018. Trimbos Instituut/Vilans/Movisie/NCJ/NISB/NJi/RIVM
- [Result] Schijven EP, VanDerNagel JEL, Otten R, Lammers J, Poelen EAP. Take it personal! Development and modelling study of an indicated prevention programme for substance use in adolescents and young adults with mild intellectual disabilities and borderline intellectual functioning. J Appl Res Intellect Disabil. 2021 Jan;34(1):307-315. doi: 10.1111/jar.12808. Epub 2020 Sep 29. PMID 32990417
- [Result] Schijven EP, Hulsmans DHG, VanDerNagel JEL, Lammers J, Otten R, Poelen EAP. The effectiveness of an indicated prevention programme for substance use in individuals with mild intellectual disabilities and borderline intellectual functioning: results of a quasi-experimental study. Addiction. 2021 Feb;116(2):373-381. doi: 10.1111/add.15156. Epub 2020 Sep 21. PMID 32678489